CLINICAL TRIAL: NCT06192459
Title: Effect of the Muscle Strength and Range of Motion Training for Post-platelet Rich Plasma Injection in People With Rotator Cuff Partial Tear: a Randomized, Cross-over Trial
Brief Title: Effect of the Muscle Strength and Range of Motion Training for Post-platelet Rich Plasma Injection in People With Rotator Cuff Partial Tear
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Hospital, Ministry of Health and Welfare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 202316
Record Dates: First submitted 2023-10-06; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Rotator Cuff Tears
Keywords: PRP; Shoulder joint mobility
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Physical Therapy Modalities; Psychotherapy, Multiple

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modality physical therapy vs combined therapy (Experimental): Participants in this are will receive one month of modality physical therapy followed by one month of modality therapy combined muscle strengthening and joint mobility training.
  Interventions: Device: Modality physical therapy; Other: Combined therapy:
- Combined therapy vs modality physical therapy (Experimental): Participants in this are will receive one month of modality therapy combined muscle strengthening and joint mobility training followed by one month of modality physical therapy.
  Interventions: Device: Modality physical therapy; Other: Combined therapy:

INTERVENTIONS:
Device: Modality physical therapy — Magnetotherapy, low-energy laser, electrotherapy, etc.
Other: Combined therapy: — Muscle strength and joint mobility training, provided twice a week for a duration of three weeks (with assessment on the second session of the third week), totaling six rehabilitation sessions. Additionally, patients are required to engage in daily home-based rehabilitation. During the hospital-based training sessions, a therapist provides guidance and conducts the training. This process encompasses progressive muscle strength training, manual joint mobilization, and active and passive joint movement training to achieve effective rehabilitation outcomes. Each rehabilitation session in the hospital lasts approximately 30 minutes. For home-based training, patients must follow the therapist's instructions and complete 20-30 minutes of home rehabilitation every day. Modality physical therapy are are carry out as usual.

SUMMARY:
Background:

Although it is known that Platelet-Rich Plasma injections have a remarkable pain relief effect for patients with partial tears of the rotator cuff in the shoulder joint, many patients still experience limited muscle strength and joint mobility recovery. Patients often inquire about post-Platelet-Rich Plasma injection rehabilitation and precautions. Therefore, it is necessary to design a comprehensive post-injection rehabilitation and training plan to improve the quality of treatment. However, previous literature on post-Platelet-Rich Plasma injection treatment seems to have inconsistent rehabilitation plans. One major reason for this inconsistency might be the lack of sufficient evidence or unclear rehabilitation effectiveness, leading to poor patient compliance. The underlying cause of these issues is the absence of a standardized and effective rehabilitation plan. Hence, it is essential to develop a standardized rehabilitation plan to enhance treatment effectiveness.

Method:

The investigators designed a non-blinded, randomized, crossover trial to observe the potential benefits of muscle strength and joint mobility rehabilitation intervention one month after PRP injection treatment for patients with partial tears of the rotator cuff. Patients were randomly divided into two groups. One group received only standard physical therapy (magneto-therapy, low-energy laser, electrotherapy, etc.), while the other group underwent muscle strength and joint mobility training in addition to standard physical therapy. There were three assessment time points: pre-assessment (one week after Platelet-Rich Plasma injection), after the first stage of treatment (three weeks of rehabilitation training + standard physical therapy/standard physical therapy following the first Platelet-Rich Plasma injection treatment), and after the second stage of treatment (three weeks of rehabilitation training + standard physical therapy/standard physical therapy following the second Platelet-Rich Plasma injection treatment).

The assessment methods included quantifying muscle strength using a hand-held dynamometer (Manual Muscle Test) and measuring three shoulder joint angles (abduction, external rotation, internal rotation). The Shoulder Pain and Disability Index recorded changes and progress in each value at different treatment stages.

Analysis: A repeated-measures Analysis of Variance model was used to analyze the trial's effects and correlations. We also analyzed whether the dose-effect existed concerning the use of time/frequency.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with rotator cuff tears who have undergone PRP (Platelet-Rich Plasma) treatment. All participants must sign an informed consent form.
2. Patients must fully participate in the rehabilitation treatment throughout the study.

Exclusion Criteria:

1. Patients with concomitant other skeletal joint issues, such as multiple joint arthritis, humeral or acromioclavicular joint fractures, or those who have undergone previous shoulder joint surgeries.
2. Patients with severe shoulder joint immobility or contracture preventing any joint movement, but mild to moderate joint mobility restrictions are not considered exclusion criteria.
3. Inability to comply with the two-month research project.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-06-11 (Estimated); Study Completion 2024-09-11 (Estimated)

PRIMARY OUTCOMES:
Manual muscle testing | pre-intervention/ three weeks after (post-first intervention)/ six weeks after (post-second intervention)
  Manual muscle testing with hand-held dynamometry.
Shoulder joint range of motion test | pre-intervention/ three weeks after (post-first intervention)/ six weeks after (post-second intervention)
  Shoulder joint range of motion test with hand-held goniometer
Shoulder Pain and Disability Index | pre-intervention/ three weeks after (post-first intervention)/ six weeks after (post-second intervention)
  self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities. The pain dimension consists of five questions regarding the severity of an individual's pain. Functional activities are assessed with eight questions designed to measure the degree of difficulty an individual has with various activities of daily living that require upper-extremity use.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Hospital, Ministry of Health and Welfare, New Taipei City, ROC, Taiwan

IPD SHARING:
Plan to Share IPD: No